CLINICAL TRIAL: NCT06355193
Title: The Use of Isatidis Root and Forsythia Oral Liquid for the Treatment of Mild Cases of COVID-19: A Trial Clinical Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Mi Zhou, Investigator, Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MZhou
Record Dates: First submitted 2024-04-08; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Treatment of Mild Cases of COVID-19
MeSH Terms: interventions — lianhuaqingwen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LGLQ group (Experimental)
  Interventions: Drug: Langenlianqiao
- LHQW group (Experimental)
  Interventions: Drug: LianhuaQingWen
- placebo control group (Placebo Comparator)
  Interventions: Other: placebo control group

INTERVENTIONS:
Drug: Langenlianqiao — The data of patients with COVID-19 mild disease treated in our Hospital from November to December 2022 were collected, and the patients were divided into 100 cases of langenlianqiao(LGLQ) treatment group, 100 cases of LianhuaQingWen(LHQW) treatment group, and 53 cases of placebo control group according to the treatments they received, and the proportion of occurrence of major clinical symptoms, the time of symptom disappearance, and the number of days in hospitalization, and the duration of infection were compared among the three groups.
  Arms: LGLQ group
Drug: LianhuaQingWen — The data of patients with COVID-19 mild disease treated in our Hospital from November to December 2022 were collected, and the patients were divided into 100 cases of langenlianqiao(LGLQ) treatment group, 100 cases of LianhuaQingWen(LHQW) treatment group, and 53 cases of placebo control group according to the treatments they received, and the proportion of occurrence of major clinical symptoms, the time of symptom disappearance, and the number of days in hospitalization, and the duration of infection were compared among the three groups.
  Arms: LHQW group
Other: placebo control group — placebo control group
  Arms: placebo control group

SUMMARY:
This study has significant implications for research, as it provides a basis for further studies on the antiviral effects of LGLQ Oral Liquid, encouraging more extensive clinical studies in larger populations and diverse age groups to validate these findings. For medical practice, the findings suggest that LGLQ can be considered an alternative treatment option for mild cases of COVID-19, especially in managing symptoms like fatigue, potentially broadening the range of effective treatments available to healthcare practitioners. In terms of policy, the demonstrated efficacy of LGLQ could lead to its inclusion in treatment guidelines for COVID-19 and other viral infections, fostering a more integrated approach combining Western medicine and Traditional Chinese Medicine in the global fight against pandemics. The insights from this study might prompt health policymakers to reassess the potential of herbal formulations in managing and treating infectious diseases and consider them in the development of future healthcare strategies and policies.

ELIGIBILITY:
Inclusion Criteria:

* the diagnosis of SARS-Cov-2 infection confirmed by quantitative polymerase chain reaction (qPCR) test
* aged 18 years or older
* patients received more than 2 doses of SARS-Cov-2 vaccine
* asymptomatic or mild at the time of hospitalization

Exclusion Criteria:

* patients with malignant diseases, autoimmune diseases, liver and kidney diseases, blood diseases, neurological diseases, endocrine diseases and other serious diseases may affect the patient's participation in the trial or affect the results of the study
* pregnant women, lactating mothers; allergic conditions
* allergic to the known components of the drug
* patients vaccinated with vaccines less than 1 shot
* Patient does not agree to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Treatment and symptomatic improvement effects of LGLQ | 1 month
  LGLQ and LHQW were able to significantly reduce the duration of infection with novel coronaviruses

CONTACTS AND LOCATIONS:
Locations (1):
- Changde Hospital, Changde, Hunan, China